CLINICAL TRIAL: NCT02808962
Title: In Pursuit of the Optimal Performance of Radiofrequency Ablation of the Nerves Supplying the Posterior Sacroiliac Joint Complex.
Brief Title: Optimal Performance of RFA of the Nerves Supplying the Posterior Sacroiliac Joint Complex.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Yakov Vorobeychik, Professor of Anesthesia, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002420
Record Dates: First submitted 2016-05-23; First posted 2016-06-22 (Estimated); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Osteoarthritis Nos, of Sacroiliac Joint
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cooled Radiofrequency Ablation (Other): This is a single arm, prospective observational study. All subjects enrolled are patients that meet the inclusion criteria, as deemed by a physician.
  Typical standard of care for these patients is an initial visit followed by two diagnostic blocks ((0.5ml) of 1% Lidocaine per level). Subjects are asked to complete the pain diary and if they experience a 75% or more decrease in the NRS, they are scheduled for Cooled RFA of the lateral branches of S1, S2, and S3 dorsal rami nerves and of the dorsal ramus of L5 nerve.
  Interventions: Procedure: Cooled RFA of sacral lateral branches

INTERVENTIONS:
Procedure: Cooled RFA of sacral lateral branches — A single target will be identified at the junction of the sacral ala and S1 superior articular process, corresponding to the location of the L5 dorsal ramus. Then, utilizing a stainless steel Epsilon Ruler (Kimberly Clark, Irving, TX, USA), three targets will be localized 8-10 mm lateral to the S1 and S2 posterior sacral foramen at the 2:30, 4:00, and 5:30 positions. Two targets will be localized at the S3 level. Local infiltration with 1% lidocaine and minimal sedation with IV midazolam will be utilized. Once suitable sensory and motor stimulation are verified and impedance is acceptable, each target will be anesthetized with 1 mL of 1% lidocaine prior to each lesion being created at 60 degrees centigrade for 2 minutes and 30 seconds.

SUMMARY:
The procedure is supposed to ablate the sacral lateral branches that form the medial cluneal nerves (MCN). The anatomy of the sacral lateral branches is such that, in addition to innervating the SIJ, distal branches of these nerves also innervate the skin over the buttock through MCN (12,13). SLB blocks (usually with 0.5 ml of 1% Lidocaine or 0.5% Bupivacaine) are performed proximal to the origin of both the nerves to the SIJ and the cutaneous branches. Therefore, a technically accurate block should anesthetize not only the SIJ but also the skin of the buttock regardless of the patient symptoms. Hypoesthesia of the buttock would, therefore, be a quality-assurance sign that the block has been performed in a technically correct fashion. Similarly, if the target nerves have been accurately ablated by RFA hypoesthesia of the buttock should ensue, as an expected effect of the procedure.

DETAILED DESCRIPTION:
Typical standard of care for these patients is initial visit followed by two diagnostic blocks ((0.5 ml) of 1 % Lidocaine per level). They are asked to complete the pain diary and if they experience a 75% or more decrease in the NRS, they are scheduled for Cooled RFA of the lateral branches of S1, S2, and S3 dorsal rami nerves and of the dorsal ramus of L5 nerve.

If patients do not experience adequate pain relief after either of these injections, it is determined that the cooled RFA procedure will not work for them. Therefore, if they fail to receive adequate pain relief after either of these two injections, they will exit the study and other alternatives will be explored. The patient will also exit the study if they fail to achieve success 1 month after RFA treatment. The treatment of the study patients will not deviate from the standard of care.

* All study Patients

  * Visit 1 - Initial Visit During the initial visit, the eligible patients will undergo a routine physical examination where it will be determined if the subject is eligible for the study. If eligible, the physician will explain the study and determine if subject is interested. Informed consent will then be obtained and the patient will be scheduled for the first fluoroscopy-guided diagnostic block with 0.5 ml of 1% Lidocaine of the lateral branches of S1, S2, and S3 dorsal rami nerves and of the dorsal ramus of the L5 nerve. The baseline information, including a 3-day average Numeric Rating Scale (NRS) regarding level of pain, the Oswestry Disability Index (ODI), and analgesic consumption will also be obtained during the initial visit.
  * Visit 2 - First Diagnostic Block The participant will be asked questions about their level of pain (NRS) and any change in analgesia medications since their last visit. They will then undergo the first fluoroscopy-guided diagnostic block (DB) with 0.5 ml of 1 % Lidocaine per level. A brief physical examination - including a sensory exam of the buttock area - will be performed after the block and the patients will be given a pain diary to complete after the procedure until the pain intensity reaches pre-procedure intensity (see the flowchart attached). The results of the exam will be documented, i.e ; "no sensory deficit" or "sensory deficit to pinprick in the buttock area". Pain diary will require the patients to scale their pain intensity using the NRS on an hourly basis and to document their activities during this period time. This will be done in accordance with the International Spine Intervention Society practice guidelines with respect to the diagnostic blocks as a prerequisite for radiofrequency ablation. (14). A follow-up appointment will be scheduled in 3-5 days after the first set of diagnostic blocks (this appointment will be pre-scheduled in conjunction with the appointment for the first diagnostic block).
  * Visit 3 - First Follow-up (3-5 days after first block) The patient will be evaluated, including NRS and analgesia medications, and the pain diary reviewed. If a 75% or more decrease in the NRS is reported for ≥ 2 hours after the procedure, the patient will be scheduled for a second set of fluoroscopy-guided diagnostic blocks (see Module 1). According to the International Spine Intervention Society and most of the major insurers' guidelines, two "positive"diagnostic blocks are necessary in order to proceed to RFA. If the first diagnostic block doesn't provide temporary ≥ 75% pain relief, the patient will exit the study.
  * Visit 4 - Confirmatory Block The participant will be asked questions about their level of pain (NRS) and any change in analgesia medications since their last visit. They will then undergo the second fluoroscopy-guided diagnostic block with 0.5 ml of 1 % Lidocaine per A brief physical examination - including a sensory exam of the buttock area - will be performed after the block and the patients will be given a pain diary to complete after the procedure until the pain intensity reaches the baseline (see the attached flowchart). The results of the sensory exam will be documented, i.e ; "no sensory deficit" or "sensory deficit to pinprick in the buttock area". This will be done in accordance with the International Spine Intervention Society practice guidelines with respect to the diagnostic blocks as a prerequisite for radiofrequency ablation. (14). A follow-up appointment will be scheduled in 3-5 days after the second set of diagnostic blocks (this appointment will be pre-scheduled in conjunction with the appointment for the second diagnostic block).
  * Visit 5 - Second Follow-up (3-5 days after 2nd block) The patients will be evaluated again at their second follow-up appointment, including NRS and analgesia medications, and the pain diary reviewed. If this block is "negative," the patient will exit the study after the follow-up and will be treated by alternative methods; if it is "positive", the patient will be scheduled for a Cooled RFA.
  * Visit 6 - Cooled RFA These subjects that experienced a "positive" response to two sets of diagnostic blocks will undergo Cooled RFA of the lateral branches of S1, S2, and S3 dorsal rami nerves and of the dorsal ramus of L5 nerve as described by Kapural et al. (15). All patients will be evaluated for buttock hypoesthesia immediately after the intervention.
  * Visit 7 - 1 Month Follow-up after Cooled RFA At this time, the following data will be collected: 3-day average NRS scores, satisfaction with the treatment, ODI, and analgesic consumption. Physical evaluation, including sensory exam of the buttock area will be done. If the procedure is successful (NRS scores improvement by ≥ 50% and satisfaction with the treatment) the patients will be scheduled for the second and final follow-up at 6 months post-intervention. Otherwise, they will exit the study.
  * Visit 8 (Final) - 6 Month Follow-up after Cooled RFA At this time, the following data will be collected: 3-day average NRS scores, satisfaction with the treatment, ODI, and analgesic consumption. Physical evaluation, including sensory exam of the buttock area will be done.
* Data to be collected The following data will be collected for each patient: Name, MRN, date of visit, NRS scores, ODI information, concomitant meds, pain diary, treatment satisfaction, and sensory exam info.

ELIGIBILITY:
Inclusion Criteria:

1. Predominantly axial pain below the L5 vertebrae
2. Pain duration of ≥ 6 months
3. Three day average NRS scores of ≥ 3/10
4. Age greater than 18 years
5. Failure of conservative treatment including nonsteroidal anti-inflammatory medications and physical therapy
6. Pain localized in the SIJ region
7. Failure of injection of steroids into the SIJ or sacroiliac ligaments to achieve adequate improvement -

Exclusion Criteria:

1. Radicular pain
2. Systemic infection or localized infection at the anticipated introducer entry site
3. Pregnancy
4. Allergy to Lidocaine
5. Individuals unable to consent
6. Bleeding dyscrasias
7. Non-English speaking patients
8. Patients that cannot read or write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02-17 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Absence/ presence of post-procedural buttock hypoesthesia | 6 months postprocedure

SECONDARY OUTCOMES:
Numeric pain rating scale (0-10) | 6-month postprocedure
Oswestry Disability Index (ODI) | 6-month postprocedure
Analgesic consumption | 6-month postprocedure
Patient satisfaction with the treatment? | 6-month postprocedure
  Binary "Yes" or "No" answer.

CONTACTS AND LOCATIONS:
Overall Officials: Yakov Vorobeychik, Principal Investigator — Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1.Patel, Gross, Brown, et al. A randomized,placebo-controlled study to assess the efficacy of lateral branch neurotomy for chronic sacroiliac joint pain. Pain Med 2012;13:383-98. 3.Tubbs, Levin, Loukas, et al. Anatomy and landmarks for the superior and middle cluneal nerves: Application to posterior iliac crest harvest and entrapment syndromes. J Neurosurg Spine 2010;13:356-569. 4 Roberts S, Burnham R, Ravichandiran K, et al. Cadaveric study of sacroiliac joint innervation: implications for diagnostic blocks and radiofrequency ablation. Regional Anesthesia and Pain Madicine 2014; 39:1-9 5. Bogduk N. (ed). Practice Guidelines for Spinal Diagnostic and Treatment Procedures, 2nd edn. International Spine Intervention Society, San Francisco, 2013 6. Kapural, Stojanovic, Bensitel. et al. Cooled Radiofrequency (RF) of L5 dorsal ramus for RF denervation of the sacroiliac joint: technical report. Pain Med. 2010; 11:53-7